CLINICAL TRIAL: NCT07353125
Title: Evaluation of the Blood Glucose Monitoring System LS-9 of Leison Biotech Co., Ltd. in Accordance With DIN EN ISO 15197:2015
Brief Title: System Accuracy and Performance Evaluation by the User of BGM LS-9
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut fur Diabetes Karlsburg GmbH (Other)
Responsible Party: Principal Investigator, Matthes Kenning, Eckhard Salzsieder, Principal Investigator, Institut fur Diabetes Karlsburg GmbH
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2025_004
Record Dates: First submitted 2026-01-06; First posted 2026-01-20 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Diabetes
Keywords: System Accuracy; Performance Evaluation by the User; DIN EN ISO 15197
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subject glucometer measurement (Experimental)
  Interventions: Diagnostic Test: Glucometer Test

INTERVENTIONS:
Diagnostic Test: Glucometer Test — blood glucose measurement using finger tip capillary blood using BGM and reference method

SUMMARY:
This study assesses the system accuracy and performance evaluation by the user of a blood glucose monitoring system pursuant to ISO 15197

ELIGIBILITY:
Inclusion criteria:

* Male or female patients with hypo-, eu- or hyperglycaemia
* The written informed consent had to be signed
* The volunteers must be older than 18 years
* The volunteers have legal capacity and are able to understand meaning, nature and possible consequences of the procedures involved

Exclusion criteria:

* Pregnancy or lactation
* Acute or chronic diseases with the risk of aggravation by the measure
* A current constitution that does not allow participating in the study
* Participation in another study or activity with the blood glucose measuring system evaluated in the present study
* Application of substances listed in Appendix A of DIN EN ISO 15197:2015

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2025-07-21 (Actual); Primary Completion 2025-09-16 (Actual); Study Completion 2025-09-22 (Actual)

PRIMARY OUTCOMES:
Analysis of system accuracy based on DIN EN ISO 15197 | Day 1
  Assessment of the analytical measurement performance of the blood glucose monitor in accordance with DIN EN ISO 15197, section 6.3
Analysis of system accuracy based on DIN EN ISO 15197 | Day 1
  Assessment of the analytical measurement performance of the blood glucose monitor in accordance with DIN EN ISO 15197, section 8

CONTACTS AND LOCATIONS:
Overall Officials: Eckhard Salzsieder, PhD, Study Director — Institut fur Diabetes Karlsburg GmbH
Locations (1):
- Institut für Diabetes Karlsburg GmbH, Karlsburg, Mecklenburg-Vorpommern, Germany

IPD SHARING:
Plan to Share IPD: No